CLINICAL TRIAL: NCT05505487
Title: Construction and Effect Evaluation of Integrated Care Model for Pulmonary Infection in Stroke Patients With Tracheotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20220324004-FS01
Record Dates: First submitted 2022-05-14; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Pulmonary Infection
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This study is a quasi-experimental study; no equal control design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Implement routine nursing such as: routine oral nursing, tracheostomy, dressing change, sputum suction nursing, oral education, etc.
- intervention group (Experimental): Implement comprehensive nursing models such as: admission risk assessment, personalized oral care based on beck oral score, aspiration prevention, airway care, diversified health education
  Interventions: Other: integrated care model

INTERVENTIONS:
Other: integrated care model — The interventions in this study were to implement basic patient care only and did not involve any invasive procedures. On the basis of routine nursing, the content of nursing intervention was integrated, and a standardized nursing model was formed for clinical application to control the severity of pulmonary infection in patients with simple tracheotomy in the non-acute phase of stroke.
  Arms: intervention group

SUMMARY:
1. To understand the occurrence of pulmonary infection in stroke patients with tracheotomy, and to clarify the current situation of clinical nursing.
2. Construct a standardized, systematic and scientific integrated care model to control the severity of pulmonary infection in non-acute stroke patients with simple tracheotomy.
3. To evaluate the clinical application effect of integrated care model of pulmonary infection in stroke patients with tracheotomy.

DETAILED DESCRIPTION:
1. Research content This study involves two parts: construction and effect evaluation.

1. The construction link includes: retrospective analysis of patient data, clinical observation, literature review, expert consultation, and pre-experiment.
2. Effect evaluation: The integrated care model was applied to the clinic, and the patients' CPIS score, Beck oral score, ZBI caregiver burden score, EQ-5D score and hospitalization cost were collected to evaluate the effect of the model.

2. The grouping method Convenience sampling method was used to select patients with simple tracheotomy for non-acute stroke who were admitted to the Department of Rehabilitation Medicine of Shenzhen Second People's Hospital as the research object, and the patients before the implementation of the integrated care model(May-July 2022) were set as the control group , the patients after the implementation of the integrated care model (August-October 2022) were set as the intervention group.

3. Sample Size Estimation

1. This study is a quasi-experimental study, and the main outcome indicator is the control of pulmonary infection (CPIS score). Therefore, the sample size estimation method of the group design quantitative data sample mean is adopted.
2. Based on the results reported in similar research literature, the authors assumed that the CPIS scores of the control group and the intervention group were 3.9±1.5 and 2.8±1.1, respectively. Set β=0.1, power (Power=1-β)=90%, two-sided α=0.05 at the significance level, and the sample size of each group was 32 cases after calculation by G-power3.1 software. According to the 20% dropout rate, the final sample size of each group was 40 cases, and there were 80 cases in the two groups.

4. Statistical analysis Using Excel and IBM SPSS Statistics 26.0 software for double entry and analysis, the measurement data that conformed to the normal distribution were expressed as the mean ± standard deviation, and the t test was used for comparison between groups; the measurement data that did not conform to the normal distribution were expressed as the median and four The number of quantiles was expressed, and the rank-sum test was used for comparison between groups. The count data were expressed as frequency and percentage, and the chi-square test was used for comparison between groups. The difference was statistically significant with p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Non-acute stroke patients diagnosed by MRI or CT who meet the diagnostic criteria of the "Chinese Guidelines for the Prevention and Treatment of Cerebrovascular Diseases";
* Those who meet the diagnostic criteria for pulmonary infection;
* Age ≥18 years old;
* Tracheotomy patients who have been off the ventilator or do not need mechanical ventilation;
* Patients who can cooperate with the research and sign the informed consent.

Exclusion Criteria:

* Patients whose vital signs are unstable and may be transferred to ICU for treatment in the future;
* Patients with malignant tumors or other infectious diseases.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-07 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Clinical Pulmonary Infection Score | Within 1 week of admission
  The scale mainly includes 7 indicators of body temperature, white blood cell count, tracheal secretions, oxygenation, chest X-ray, progress of pulmonary exudation, and microbial culture of tracheal aspirates, each with 0 to 2 points, with a total score of 12 If the score is less than 6, the lung infection is considered to be controlled.
Clinical Pulmonary Infection Score | 3 weeks after admission
  The scale mainly includes 7 indicators of body temperature, white blood cell count, tracheal secretions, oxygenation, chest X-ray, progress of pulmonary exudation, and microbial culture of tracheal aspirates, each with 0 to 2 points, with a total score of 12 If the score is less than 6, the lung infection is considered to be controlled.

SECONDARY OUTCOMES:
Beck Oral Assessment Score(BOAS)，modified | Within 1 week of admission
  The scale includes five items: lips, gums and oral mucosa, tongue, teeth, and saliva to evaluate the oral hygiene status and functional status. Each item is scored with 1 to 4 points, and the total oral hygiene score is 5 to 20 points. The higher the score, the worse the oral hygiene.
Beck Oral Assessment Score(BOAS)，modified | 3 weeks after admission
  The scale includes five items: lips, gums and oral mucosa, tongue, teeth, and saliva to evaluate the oral hygiene status and functional status. Each item is scored with 1 to 4 points, and the total oral hygiene score is 5 to 20 points. The higher the score, the worse the oral hygiene.
Zarit Caregiver Burden Interview, ZBI | Within 1 week of admission
  The scale mainly includes 2 dimensions (personal burden and responsibility burden), a total of 22 items, each item is divided into 5 grades according to the severity of the burden, expressed on a scale of 0-4, 0 means never, 4 means almost often. The total score of the scale is 0-88 points, and the higher the score, the heavier the burden of care.
Zarit Caregiver Burden Interview, ZBI | 3 weeks after admission
  The scale mainly includes 2 dimensions (personal burden and responsibility burden), a total of 22 items, each item is divided into 5 grades according to the severity of the burden, expressed on a scale of 0-4, 0 means never, 4 means almost often. The total score of the scale is 0-88 points, and the higher the score, the heavier the burden of care.
EuroQol-5 Dimension， EQ-5D | Within 1 week of admission
  he Chinese version of the European five-dimensional health scale (EuroQol-5 Dimension, EQ-5D), EQ-5D is a commonly used scale to measure health-related quality of life. The scale is divided into 2 parts: the EQ-5D health description system and the EuroQol-Visual Analogue Score (EQ-VAS). The EQ-5D health description system includes 5 dimensions: mobility, self-care, activities of daily living, pain or discomfort, anxiety or depression, and each dimension contains 3 levels: no difficulty, some difficulty, and extreme difficulty. The EQ-VAS uses a score of 0 to 100 to evaluate a patient's current health status, with 100 representing the "best health status in my mind" and 0 representing the "worst health status in my mind".
EuroQol-5 Dimension， EQ-5D | 3 weeks after admission
  he Chinese version of the European five-dimensional health scale (EuroQol-5 Dimension, EQ-5D), EQ-5D is a commonly used scale to measure health-related quality of life. The scale is divided into 2 parts: the EQ-5D health description system and the EuroQol-Visual Analogue Score (EQ-VAS). The EQ-5D health description system includes 5 dimensions: mobility, self-care, activities of daily living, pain or discomfort, anxiety or depression, and each dimension contains 3 levels: no difficulty, some difficulty, and extreme difficulty. The EQ-VAS uses a score of 0 to 100 to evaluate a patient's current health status, with 100 representing the "best health status in my mind" and 0 representing the "worst health status in my mind".

OTHER OUTCOMES:
hospital costs | ≥3 weeks
  Collection of treatment expenses during hospitalization of patients through the hospital electronic medical record system

CONTACTS AND LOCATIONS:
Overall Officials: Yan Gao, Ph.D, Principal Investigator — Shenzhen Second People's Hospital
Locations (1):
- The Second People's Hospital of Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Contact the principal investigator for data if necessary